CLINICAL TRIAL: NCT00601198
Title: Phase II Study of the Efficacy of Amifostine (Ethyol) in Reducing the Incidence and Severity of Oxaliplatin-Induced Neuropathy in Patients With Colorectal Cancer
Brief Title: A Study of Amifostine (Ethyol) in Patients With Colorectal Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Funding support withdrawn
Sponsor: University of Cincinnati (Other)
Collaborators: MedImmune LLC (Industry); AstraZeneca (Industry)
Responsible Party: Principal Investigator, Michelle Marcum, Director of University of Cincinnati Cancer Center, University of Cincinnati
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ETH190-06; ETH190-06
Record Dates: First submitted 2008-01-14; First posted 2008-01-25 (Estimated); Results first posted 2023-08-01 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Colorectal Cancer
Keywords: Oxaliplatin-induced Neuropathy; Colon and rectum
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Amifostine; Fluorouracil; Leucovorin; Oxaliplatin; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment Period (Experimental): The chemotherapy regimen will be given for 2 consecutive days. On day #1, pt. will be premedicated with drugs to prevent nausea and vomiting in addition to intravenous fluids. Then they will receive amifostine intravenously followed by oxaliplatin, 5FU and leucovorin. This will be followed by an infusion of 5FU given in a pump over 22 hours. If the doctor decides on giving the pt. Avastin, this will be given on day #1. On day #2, they will receive the same treatment except for oxaliplatin.
  Interventions: Drug: Amifostine

INTERVENTIONS:
Drug: Amifostine — Patients should be treated with oxaliplatin-based chemotherapy in combination with amifostine for 12 cycles, or until unacceptable toxicity is observed or disease progression
  Other Names: Flurouracil (5-FU); Leucovorin calcium (LV); Oxaliplatin; Bevacizumab

SUMMARY:
The purpose of this study is to determine the effect of amifostine (ETHYOL) on decreasing the rate and severity of nerve dysfunction or neuropathy (numbness and tingling in hands and feet) associated with FOLFOX chemotherapy.

DETAILED DESCRIPTION:
In addition, this study will provide information on how subjects with colorectal cancer do while receiving amifostine in combination with other chemotherapy drugs. This study will also look at the frequency of complications associated with amifostine and chemotherapy.

The FOLFOX chemotherapy regimen consists of three drugs, 5-FU, leucovorin, and oxaliplatin, all given intravenously (into the vein) every 2 weeks with or without Avastin given in combination with chemotherapy. FOLFOX has been approved by the Food and Drug Administration (FDA) for the treatment of cancer of the colon or rectum.

Amifostine is not a chemotherapy drug. It is approved by the Food and Drug Administration (FDA) to prevent moderate or severe dryness of the mouth caused by radiation treatment for head and neck cancer, and to prevent kidney damage caused by cisplatin chemotherapy treatment for ovarian and non-small cell lung cancer. Amifostine is not FDA approved for use in this study and is therefore considered investigational.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically-proven adenocarcinoma of the colon or rectum
* AJCC stage II, III or IV
* Male of female aged greater than or equal to 18 years
* ECOG Performance Status (PS): 0-2
* Men or women of reproductive potential must have agreed to use an effective method of contraception while on treatment and for 6 months after study treatment
* If female, not pregnant or lactating. Documentation of a negative serum HCG pregnancy test for women of childbearing potential is required within 7 days prior to be considered of non-childbearing potential
* In the opinion of the investigator, patients must have a life expectancy of least 6 months
* At the time of study enrollment, absolute granulocyte count (AGC) must be greater than or equal to 1500/mm3, platelet count must be greater than or equal to 100,000/mm3
* There must be evidence of adequate hepatic and renal function. Bilirubin less than or equal to UNL, Alkaline phosphatase less than or equal to 2.5xULN, AST less than or equal to 1.5xULN, Creatine less than or equal to 1.5xULN
* Signed written informed consent obtained prior to study-specific screening procedure

Exclusion Criteria:

* Any condition or past medical history that contra-indicate treatment with oxaliplatin and 5FU, as reported in the approval labeling information
* Hypersensitivity to any of the study treatments (amifostine, oxaliplatin and 5FU) or ingredients
* Received any investigational drug within 30 days before beginning treatment with study drug
* Concomitant treatment with other investigational agents
* Received prior oxaliplatin or cisplatin based chemotherapy
* History of peripheral neuropathy
* concomitant treatments with drugs/ingredients reported to have a potential activity in preventing peripheral sensory neuropathy: carbamazepine, gabapentin, phenytoin, gluthathione, alpha-lipoic acid, celecoxib, venlafaxine, vitamin B1 (thiamine), B6 (pyridoxine), ginko biloba. Multivitamins and dietary supplements are allowed. Uncontrolled intercurrent illness: e.g. high blood pressure, unstable angina, symptomatic congestive hear failure (NY Heart Association Classification III or IV), serious cardiac arrhythmia, diabetes, or active infection
* Concurrent active cancer originating from a primary site other than colon or rectum
* Presence of any symptom suggesting brain/spinal cord metastasis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2006-10; Primary Completion 2010-01-13 (Actual); Study Completion 2010-01-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Marcum, Study Director — University of Cincinnati
Locations (1):
- University of Cincinnati, Cincinnati, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment Period
Started | 4
Completed | 4
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment Period
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 50.83 [45.09 to 56.02]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 2
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 2
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 4

OUTCOME MEASURES:

1. Primary Outcome: Test Drug in 28 Patients and Assess PSN. If 5 or More Have Grade 3 & 4 PSN, Trial Will be Terminated.
Description: There were only four participants in this study. None of which completed the questionnaires needed to assess this outcome. This study was closed by the sponsor on January 13, 2010 due to low enrollment.
Time Frame: 2 years
Population: There were only four participants in this study. None of which completed the questionnaires needed to assess this outcome. This study was closed by the sponsor on January 13, 2010 due to low enrollment.
Arm/Group | Treatment Period
Number analyzed (Participants) | 0

2. Secondary Outcome: Assess PSN in 69 Patients. If Total Number of Cumulative PSN is > or Equal to 14, Drug Will be Rejected.
Description: as for outcome 1
Time Frame: 1 year
Population: as for outcome 1
Arm/Group | Treatment Period
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Treatment Period
All-Cause Mortality (participants affected / at risk) | 1/4
Serious Adverse Events (participants affected / at risk) | 2/4
Other Adverse Events (participants affected / at risk) | 2/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Period (N=4)
Small bowel obstruction (Gastrointestinal disorders) | 1 (1)
Dehydration (Gastrointestinal disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
Leukocytosis (Investigations) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Period (N=4)
Visual changes (Eye disorders) | 1 (1)
Abnormal pain (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 2 (2)
Gum problems (Gastrointestinal disorders) | 1 (1)
Mucositis (Gastrointestinal disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 2 (2)
Taste alteration (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2)
Bone pain (General disorders) | 1 (1)
Edema limbs (General disorders) | 1 (1)
Fatigue (General disorders) | 2 (2)
Pain (General disorders) | 1 (1)
Hand foot skin reaction (Immune system disorders) | 1 (1)
Oral thrush (Infections and infestations) | 1 (1)
Albumin- low (Investigations) | 1 (1)
Alkaline phosphatase low (Investigations) | 1 (1)
ANC - low (Investigations) | 1 (1)
AST level (Investigations) | 1 (1)
Hemoglobin- low (Investigations) | 1 (1)
INR-high (Investigations) | 1 (1)
Platelet - low (Investigations) | 2 (4)
Sodium - low (Investigations) | 2 (2)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (2)
Jaw problem (Musculoskeletal and connective tissue disorders) | 1 (1)
Lumbar Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Hyperactivity (Nervous system disorders) | 1 (1)
Neuropathy (Nervous system disorders) | 2 (2)
Tingling in lip (Nervous system disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1)
Hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritis (Skin and subcutaneous tissue disorders) | 1 (1)
Flushing (Vascular disorders) | 1 (1)
Hot flashes (Vascular disorders) | 1 (1)
Warmth (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No